CLINICAL TRIAL: NCT06778837
Title: Validation of Wearable Sensors to Monitor Tissue Hydration and Stiffness in Patients With Lymphedema
Brief Title: Lymphedema Sensor Technology Development Study
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Principal Investigator, Ann Marie Flores, Associate Professor at Northwestern University, Department of Physical Therapy and Human Movement Sciences, Director of Cancer Rehabilitation Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Director of Cancer Rehabilitation Stud, Northwestern University
Other Study IDs: STU00222670
Record Dates: First submitted 2025-01-02; First posted 2025-01-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Lymphedema Arm; Lymphedema; Cancer
Keywords: Sensor; Device; Lymphedema; Upper Extremity; Wearable; Tissue; Hydration; Stiffness; Cancer
MeSH Terms: conditions — Lymphedema; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Participants
  Interventions: Device: Wearable devices to detect lymphedema

INTERVENTIONS:
Device: Wearable devices to detect lymphedema — All participants will undergo measurement of the upper extremities to test the validity and safety of wearable sensors to measure lymphedema.

SUMMARY:
The goal of this clinical trial in adult patients diagnosed with upper extremity lymphedema is to test the safety and effectiveness of small, wearable sensors that may be able to measure lymphedema. The main questions this study aims to answer are:

* Do these sensors detect lymphedema?
* If so, how accurate are these wearable sensors?

Participants will complete one in-person measurement session and one phone call with study staff 14 days after the measurement session to check-in on the participant's well-being.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of unilateral lymphedema that affects the upper extremity (UE).
* Patients previously diagnosed with non-metastatic cancer.
* Adults 18 years of age and older.

Exclusion Criteria:

* Patients with history of lymphatic surgery.
* Patients with implantable devices (e.g., pacemaker, pacemaker/defibrillator, intrathecal pump, joint replacements, etc.) or any other device deemed unsafe by the treating investigator.
* Patients with an amputation involving the upper extremity.
* Patients with known allergies to adhesives - including silicone adhesives.
* Patients with the following comorbidities: diabetes, congestive heart failure, peripheral vascular disease, irradiated upper extremity skin, psoriasis, atopic dermatitis, open wounds/skin breakdown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit patients using the above specified criteria in the Chicagoland area.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-14 (Actual)

PRIMARY OUTCOMES:
Tissue Hydration Score Recorded from the Tissue Hydration Sensor | From enrollment to the end of the measurement session (appx. 3 hours)
  This score will determine whether or not fluid associated with lymphedema is detected when compared to previously validated measures (bioimpedance spectroscopy and tissue dielectric constant). This is a continuous ratio level of measurement.
Tissue Stiffness Score from the Tissue Stiffness Sensor | From enrollment to the end of the measurement session (appx. 3 hours)
  This score will determine whether or not tissue affected by lymphedema can yield is detected when compared to a comparable clinical measurement device using Young's Modulus. This is a continuous ratio level of measurement.

SECONDARY OUTCOMES:
Bioimpedance spectroscopy (BIS) L-Dex score | Three hours
  The bioimpedance spectroscopy L-Dex score is a ratio that represents the difference in the amount of extracellular fluid in an at-risk limb compared to an unaffected limb.
Tissue Dielectric Constant (TDC) | From enrollment to the end of the measurement session (appx. 3 hours)
  The tissue dielectric constant (TDC) is derived from an electromagnetic wave that is reflected back from transmission into the tissue. It represents free and bound water in the tissue.
Volume of the Upper Extremities | Three hours
  Circumferential volumetric measurement is obtained by modeling the limb as a frustum and taking a series of circumferential measurements using anatomical landmarks at predetermined intervals (typically every 4cm), beginning at the wrist and ending at the anterior axillary fold. Volume differences of +10% represents the presence of lymphedema.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided